CLINICAL TRIAL: NCT00267930
Title: A Pilot Phase II, Randomised, Double-Blind, Placebo-Controlled, Multi-Centred Safety, Tolerability and Preliminary Efficacy Study of RSD1235-SR for the Prevention of Atrial Fibrillation/Atrial Flutter (AF/AFL) Recurrence in Subjects Post-Conversion Form AF
Brief Title: Study of RSD1235-SR for the Prevention of Atrial Fibrillation/Atrial Flutter Recurrence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advanz Pharma (Industry)
Responsible Party: Gregory Beatch, Ph.D., Vice President, Scientific Affairs, Cardiome Pharma Corp.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1235-SR-1005
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Atrial Fibrillation
Keywords: AFib; AF
MeSH Terms: conditions — Atrial Fibrillation | interventions — vernakalant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Tier 1: 1 placebo capsule b.i.d Tier 2: 2 placebo capsules b.i.d
  Interventions: Drug: Placebo comparator
- 2 (Experimental): Tier 1: Vernakalant (oral) 1 x 300 mg capsule b.i.d
  Interventions: Drug: Vernakalant (oral)
- 3 (Experimental): Tier 2: Vernakalant (oral) 2 x 300 mg (600 mg) b.i.d
  Interventions: Drug: Vernakalant (oral)

INTERVENTIONS:
Drug: Vernakalant (oral)
  Other Names: RSD1235-SR
  Arms: 2; 3
Drug: Placebo comparator
  Arms: 1

SUMMARY:
This study is designed to evaluate the safety, tolerability and preliminary efficacy of vernakalant (oral) in subjects with sustained atrial fibrillation of greater than 72 hours and less than 6 months duration

ELIGIBILITY:
Inclusion Criteria (partial list):

* Subjects must have sustained, symptomatic atrial fibrillation for greater than 72 hours and less than 6 months duration
* Subjects must have adequate anticoagulant therapy

Exclusion Criteria (partial list):

* Subjects may not have Class III or Class IV congestive heart failure
* Subjects may not have uncorrected electrolyte imbalance

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2005-12; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
All subjects who were exposed to the investigational medication were evaluated for safety. | Subjects were assessed for safety within Day 58 of dosing

SECONDARY OUTCOMES:
Recurrence of AF/AFL or withdrawal | Time for recurrence of AF/AFL or withdrawal within Day 28 of dosing
Improvement in AF symptoms | Time to improvement in AF symptoms within Day 28 of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Greg Beatch, PhD, Study Director — Advanz Pharma
Locations (22):
- United States (4):
  - The Heart Center, P.C., Huntsville, Alabama
  - Cardiovascular Consultants Medical Group, Inc., Walnut Creek, California
  - Penn State Heart & Vascular Institute, Hershey, Pennsylvania
  - Marshfield Clinic, Marshfield, Wisconsin
- Canada (2):
  - Foothills Hospital, Calgary, Alberta
  - Centre Hospitalier de l'Université de Montréal (CHUM) Hôtel Dieu, Montreal, Quebec
- Denmark (9):
  - Aalborg Sygehus Syd, Aalborg
  - Aarhus Sygehus Kardiologisk Afd. A, Aarhus
  - Bispebjerg Hospital, Copenhagen
  - Kardiologisk/endokrinologisk afd. E Frederiksberg Hospital, Frederiksberg
  - KAS Gentofte Kardiologisk Afdeling, Hellerup
  - KAS Herlev, Herlev
  - Sygehus Vendsyssel Hjorring, Hjørring
  - Medicinsk Afdeling Kolding Sygehus, Kolding
  - Roskilde Amts Sygehus Koge, Køge
- Netherlands (7):
  - Reinier de Graaf Gasthuis, Delft
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen (UMCG), Groningen
  - Trial sectie Cardiologie, Heerlen
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Stichting Sint Antonius Ziekenhuis, Nieuwegein

REFERENCES:
- See also: Related Info — http://www.cardiome.com